CLINICAL TRIAL: NCT02793375
Title: Does Montelukast Decrease Post Adenotonsillectomy Pain in Children? A Randomized Controlled Trial
Brief Title: Does Montelukast Decrease Post Adenotonsillectomy Pain in Children
Acronym: Montelukast
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN_Montelukast_001
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pain
Keywords: Montelukast; Tonsillectomy
MeSH Terms: conditions — Pain | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Patients receiving placebo preoperatively (blinded)
  Interventions: Drug: Placebo
- Study group (Experimental): Patients receiving montelukast preoperatively (blinded)
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — Age appropriate dose of Montelukast given to patients prior to undergoing adenotonsillectomy, and the day after surgery, with pain scores and amount of opioid pain medication required measured postoperatively.
  Arms: Study group
Drug: Placebo — Age appropriate dose of placebo given to patients prior to undergoing adenotonsillectomy, and the day after surgery, with pain scores and amount of opioid pain medication required measured postoperatively.
  Arms: Control

SUMMARY:
Objective: The purpose of the present study is to evaluate the effectiveness of preoperative Montelukast as an analgesic for adenotonsillectomy

Study Design: Randomized controlled double blinded clinical trial.

Setting: Cincinnati Children's Hospital Medical Center (CCHMC), Division of Pediatric Otolaryngology, Head and Neck Surgery

Methods: Children between the age of 3-8 undergoing adenotonsillectomy with planned 23 hour observation for adenotonsillar hypertrophy and sleep disordered breathing will be randomized to receive either montelukast or placebo in Same Day surgery.

Analysis: Differences in demographics (age, gender, race, weight) between the intervention and control groups will be assessed using chi-square (for categorical measures) and t tests (for continuous measures). Differences in postoperative opioid usage, postoperative pain scores using the FLACC scale, and the number of postoperative contacts (Emergency department visits or phone calls) with patients or their family regarding pain or tonsillar hemorrhage will be evaluated using chi-square (categorical measures) and t tests (continuous measures).

DETAILED DESCRIPTION:
Adenotonsillectomy (T&A) is the one of the most common pediatric procedures performed in the United States, with over 530,000 procedures performed annually1. Pain control after T&A is essential for improving recovery and enhancing quality of life. At CCHMC, our current protocol in patients over the age of three is to treat pain with scheduled Tylenol, ibuprofen and steroids, as well as opioids (oxycodone) as a "rescue" medication for uncontrolled pain. Despite this regimented approach, pain control is often suboptimal, and numerous doses of opioids are often required. Montelukast is a cysteinyl leukotriene receptor antagonist that may have a role in decreasing post T&A pain2. The primary objective of the present study is to evaluate the effect of montelukast on post-T&A pain by measuring the amount of opioid pain medication required postoperatively in patients receiving montelukast preoperatively compared to those receiving placebo. The secondary objective will evaluate post-surgical outcomes and include group comparisons of post T&A pain scores and number of Emergency department visits and/or phone calls for perioperative pain related complaints.

Hypothesis #1 Preoperative montelukast will decrease the amount of opioid pain mediation required in the first 24 hours postoperatively compared to those in the control group.

Hypothesis #2 Preoperative montelukast will decrease pain scores in the first 24 hours after surgery in patients undergoing T&A compared to those in the control group.

Hypothesis#3 Preoperative montelukast will decrease the number of postoperative contacts (Emergency department visits and phone calls) by parents for pain related concerns in the first 3-4 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria: All patients between the ages of 3-8 undergoing adenotonsillectomy for an indication of adenotonsillar hypertrophy who are scheduled for overnight 23 hour observation at CCHMC main campus.

Exclusion Criteria: Patients with moderate to severe developmental delay will be excluded due to difficulties in scoring postoperative pain. In addition, those with allergies to Montelukast and those currently using Montelukast will be excluded. Those with moderate to severe cardiac, hepatic, pulmonary or renal disease will be excluded. All patients with a primary indication of chronic tonsillitis will be excluded. Those with active respiratory infections requiring cancellation of surgery will be excluded based on the Anesthesia services recommendations.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Opioid amount | first 23 hours postoperatively
  Amount of opioid necessary for adequate pain control in first 23 hours after surgery.

SECONDARY OUTCOMES:
Pain scores | up to first 23 hours
  The use of the FLACC pain scale to determine what pain scores are in the PACU and in the first 23 hours after tonsillectomy.
Postoperative physician contacts | 4 weeks
  The number of physician phone calls and trips to the emergency room in the first month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro D deAlarcon, MD, MPH, Principal Investigator — Cincinnati Childrens Hospital and Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No